CLINICAL TRIAL: NCT00482898
Title: A Multicenter, Randomized, Double-Blind, Crossover Study Comparing the Effect of MK0359 and Placebo in Adult Patients With Chronic Asthma
Brief Title: A Study of MK0359 in Patients With Chronic Asthma (0359-013)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0359-013; MK0359-013; 2007_575
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0359

SUMMARY:
A study to test the effect of MK0359 in lessening the symptoms of asthma as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* You are between the ages of 18 and 45
* You have had a history for at least a year of COPD symptoms
* Your current asthma treatment is limited to short-acting beta-agonists(such as albuterol)
* You have a history of smoking one pack of cigarettes per day for 7 years
* You will not be away from home for more than 5 days during the study

Exclusion Criteria:

* You are unwilling to limit your alcohol use to less than 5 drinks per week
* You have been in a research study with an investigational drug or vaccine in the last 4 weeks
* You have donated blood in the last 4 weeks
* You have been hospitalized or had major surgery in the last 4 weeks
* You have been treated in the emergency room within the last 4 weeks or hospitalized within the last 3 months for your asthma
* You have a history of heart problems in the last 6 months
* You have a history of stomach problems
* You are unwilling to avoid grapefruit juice throughout the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2002-09; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Lu S, Liu N, Dass SB, Reiss TF, Knorr BA. Randomized, placebo-controlled study of a selective PDE4 inhibitor in the treatment of asthma. Respir Med. 2009 Mar;103(3):342-7. doi: 10.1016/j.rmed.2008.10.024. Epub 2009 Jan 8. PMID 19135348